CLINICAL TRIAL: NCT06375629
Title: A Multi-institutional Prospective Data Collection of Patients Treated With Partial Gland High-Intensity Focused Ultrasound (HIFU) Ablation for Prostate Cancer
Brief Title: ES-HIFU, Prospective Data Collection of Patients Treated With Partial Gland HIFU Ablation for Prostate Cancer
Acronym: ES-HIFU
Status: Terminated | Type: Observational
Why Stopped: The study was terminated early to integrate sites into a larger registry for a more comprehensive dataset, and not due to any safety concerns.
Sponsor: EDAP TMS S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: EDAP TMS
Record Dates: First submitted 2024-03-07; First posted 2024-04-19 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: FocalOne — The objective of this study is to evaluate the clinical effectiveness and safety of treatment of prostate cancer in patients who have received a focal HIFU treatment using the Focal One medical device. This study is a non-interventional study. All the data will be collected from routine care. Data as indicated in the table below will be systematically recorded on the e-CRF to coincide with the scheduled follow-up visits at 3, 6 and 12 months.

SUMMARY:
The objective of this study is to evaluate the clinical effectiveness and safety of treatment of prostate cancer in patients who have received a focal HIFU treatment using the Focal One medical device.

ELIGIBILITY:
Inclusion Criteria:

* Patient eligible for HIFU treatment for prostate cancer, excluding whole gland treatment.
* Patient newly diagnosed with localized prostate cancer confirmed with an image guided biopsy (MRI and/or micro-ultrasounds).
* Gleason ≤ 4+3.
* Patient scheduled for HIFU treatment as determined by the physician.
* Patient with healthcare coverage. Spanish-speaking patients with the ability to provide informed written consent

Exclusion Criteria:

* Patient with bilateral prostate cancer requiring whole gland treatment.
* Patients clinically detected metastasis.
* Patient with an extension of cancer or seminal vesicle invasion.
* Patient with contraindications for HIFU treatment: please refer to the complete Focal One user manual.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with localized prostate cancer and eligible for HIFU treatment for prostate cancer, excluding whole gland treatment.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Evaluation of adverse events | 1 year
  using the Clavien-Dindo classification
Evaluation of quality of life | 3, 6, 9 and 12 months
  IQL questionnaires
Evaluation of urinary incontinence | 3, 6, 9 and 12 months
  ICIQ questionnaire
Erectile function assessment | 3, 6, 9 and 12 months
  IIEF-5 questionnaire
Urinary Symptoms | 3, 6, 9 and 12 months
  IPSS questionnaire

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital General Universitario Gregorio Marañón C/ Doctor Esquerdo, Madrid
  - Hospital Universitario Central De Asturias, Oviedo
  - Hospital Universitario Marqués De Valdecilla, Santander
  - Hospital Consorcio General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No